CLINICAL TRIAL: NCT02023021
Title: A Phase II, Single-arm Study to Evaluate the Efficacy and Safety of the Combination of Nab-paclitaxel and Gemcitabine in Treating Patients With Pancreatic Cancer After Curative Resection
Brief Title: Nab-paclitaxel Combined With Gemcitabine as Adjuvant Therapy for Pancreatic Cancer After Curative Resection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xian-Jun Yu (Other)
Responsible Party: Sponsor-Investigator, Xian-Jun Yu, M.D., Ph.D., Fudan University
Organization: Fudan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABX-1312129-8
Record Dates: First submitted 2013-12-23; First posted 2013-12-30 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Stage IA Pancreatic Adenocarcinoma; Stage IB Pancreatic Adenocarcinoma; Stage IIA Pancreatic Adenocarcinoma; Stage IIB Pancreatic Adenocarcinoma
Keywords: Pancreatic Cancer; Pancreatic Adenocarcinoma; Nab-paclitaxel; Gemcitabine; Adjuvant Therapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- nab-paclitaxel + gemcitabine (Experimental): nab-paclitaxel at 100 mg/m^2 on days 1, 8, and 15; gemcitabine at 1000 mg/m^2 on days 1, 8, and 15
  Interventions: Drug: nab-paclitaxel; Drug: gemcitabine

INTERVENTIONS:
Drug: nab-paclitaxel — Patients firstly receive nab-paclitaxel 100 mg/m^2 (iv, 30 minutes) on days 1, 8, and 15 for 3 weeks, followed by one week without treatment. Treatment repeats every 4 weeks for up to 6 circles in the absence of disease recurrence or unacceptable toxicity.
  Other Names: Abraxane
Drug: gemcitabine — Patients secondly receive gemcitabine 1000 mg/m^2 (iv, 30 minutes) on days 1, 8, and 15 for 3 weeks, followed by one week without treatment. Treatment repeats every 4 weeks for up to 6 circles in the absence of disease recurrence or unacceptable toxicity.
  Other Names: GEMZAR

SUMMARY:
Pancreatic cancer has an extremely poor prognosis with a 5-year survival rate of less than 5%. About 25% of patients have the opportunity for radically surgical resection when diagnosis. However, the recurrence rate is up to 85% within 2 years. Data from clinical trials indicated that gemcitabine-based adjuvant chemotherapy reduced recurrence and enhanced overall survival for patients who have undergone surgery to remove their tumor. Nab-paclitaxel could enhance the intratumoral concentration of gemcitabine; recent studies showed that nab-paclitaxel plus gemcitabine significantly improved progression-free survival and overall survival of metastatic pancreatic cancer patients. The present study is intended to investigate the activity and safety of the combination of gemcitabine and nab-paclitaxel as adjuvant chemotherapy in treating patients with pancreatic cancer after curative resection.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed content obtained prior to treatment
* Age ≥ 18 years and ≤ 75 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Patients must have histologically confirmed pancreatic adenocarcinoma (or any mixed pathology if adenocarcinoma is predominant) after curative resection (R0). The pathological staging does not exceed the stage IIB.
* No tumor lesions are seen by abdominal and thoracic CT scan 4~8 weeks after surgery, and no serious adverse events are occurred during this period
* The expected survival after surgery ≥ 6 months
* White blood cell (WBC) ≥ 3 × 109/L; Absolute neutrophil count (ANC) ≥ 1.5 × 109/L; Platelets (PLT) ≥ 100 × 109/L; Hemoglobin (Hgb) ≥ 9 g/dL
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]/ alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) ≤ 2.5 × institutional upper limit of normal (ULN); Total bilirubin (TBIL) ≤ ULN; Creatinine (CRE) ≤ 1.5 × ULN
* Prothrombin time (PT) and international normalized ratio (INR) ≤ 1.5 × ULN

Exclusion Criteria:

* Active second primary malignancy or history of second primary malignancy within the last 3 years
* Patients who have received any form of anti-tumor therapy before surgery, including chemotherapy, radiotherapy, interventional chemoembolization, radiofrequency ablation, and molecular targeted therapy
* Use of any other investigational agents
* Patients with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, internal hemorrhage, pancreatic leakage, bile leakage, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* History of allergic reactions attributed to compounds of similar chemical or biological composition to nab-paclitaxel or gemcitabine
* Metabolic acidosis, acute or chronic, including ketoacidosis
* Pregnant or nursing women
* Human immunodeficiency virus (HIV)-positive patients
* Patients who are unwilling or unable to comply with study procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Recurrence-free survival at one year after curative resection | From date of enrollment (after curative resection) until the date of first documented recurrence or date of death from any cause, whichever came first, assessed 2 months during therapy and 3 months thereafter up to 24 months
  To evaluate the therapeutic efficacy of nab-paclitaxel plus gemcitabine chemotherapy in terms of recurrence-free survival in patients with pancreatic cancer at one year after curative resection. Computed tomography (CT) scan

SECONDARY OUTCOMES:
Overall survival after curative resection | From date of enrollment (after curative resection) until the date of death from any cause, assessed one month during therapy and 3 months thereafter up to 24 months
  To evaluate the overall survival of patients (after curative resection) treated with this regimen. Outpatient visit, phone interview
Quality of life score after curative resection | One month during therapy and 3 months thereafter up to 24 months
  To evaluate the quality of life score of patients (after curative resection) treated with this regimen. Outpatient visit, phone interview
Number of grade 3 and 4 toxicities according to NCI CTCAE version 4.0 | One week during therapy and 3 months thereafter up to 24 months
  To evaluate the occurrence of grade 3 and 4 toxicities according to National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE; version 4.0) in patients treated with this regimen. The toxicity profile includes but not limits neutropenia, thrombocytopenia, peripheral neuropathy, hypoglycemia, metabolic acidosis (acute or chronic, including ketoacidosis), which will be summarized as the percentage of patients by type and grade according to treatment group. Outpatient visit, laboratory findings
CA199 level after curative resection | One month during therapy and 3 months thereafter up to 24 months
  To evaluate the CA199 level of patients (after curative resection) treated with this regimen. Outpatient visit, laboratory findings

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Jun Yu, M.D., Ph.D., Principal Investigator — Department of Pancreatic Surgery, Fudan University Shanghai Cancer Center; Shanghai Pancreatic Cancer Institute; Pancreatic Cancer Institute, Fudan University. Shanghai, China.
Locations (1):
- Department of Pancreatic Surgery, Fudan University Shanghai Cancer Center; Shanghai Pancreatic Cancer Institute; Pancreatic Cancer Institute, Fudan University. Shanghai, China, Shanghai, China